CLINICAL TRIAL: NCT04505410
Title: A Randomized Control Study to Examine the Influence of a Healthy Diet on Moderate to Severe Ulcerative Colitis Patients Undergoing Second Line Induction With Advanced Therapies
Brief Title: Second Line Induction Therapy and Healthy Diet for Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Oriana Mazorra Damas, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20200436
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication plus FMD group (Experimental): Participants in this group with UC consuming a standard, regular low-fiber diet will start an advanced therapy for eight consecutive weeks with the addition of two, five-day cycles of Fast Mimicking Diet (FMD) daily meals on weeks 2 and 7.
  Interventions: Other: A plant based high fiber diet that mimics fasting ("FMD") plus advanced therapy
- Medication only group (Active Comparator): Participants in this group with UC consuming a diet based on tolerance will start an advanced therapy for eight consecutive weeks.
  Interventions: Drug: Advanced therapy only without dietary intervention

INTERVENTIONS:
Other: A plant based high fiber diet that mimics fasting ("FMD") plus advanced therapy — Patients will do two 5-day cycles of a fasting mimicking diet. They will start the first diet cycle 1 week after initiating a new advanced therapy: Tofacitinib and Upadacitinib (JAK inhibitors), Infliximab (anti-TNF), Ustekinumab or Risankizumab (IL-23 inhibitors).
  Arms: Medication plus FMD group
Drug: Advanced therapy only without dietary intervention — Patients in this group will start an advanced therapy and follow a diet solely based on dietary tolerance: new advanced therapy: Tofacitinib and Upadacitinib (JAK inhibitors), Infliximab (anti-TNF), Ustekinumab or Risankizumab (IL-23 inhibitors).
  Arms: Medication only group

SUMMARY:
The purpose of this study is to determine whether a diet intervention (the Fasting Mimicking diet) will help induce clinical and biochemical response to an advanced therapy in patients with ulcerative colitis. Study period will be 8 weeks during induction of advanced therapies. The primary aims of this study will be clinical response, as determined by the simple clinical colitis activity index (SCCAI). Secondary outcomes will be improvement in fecal calprotectin and C-reactive protein levels.

DETAILED DESCRIPTION:
Advanced therapies included will be:

JAK inhibitors (tofacitinib or upadacitinib) IL-23 inhibitors (ustekinumab or risankizumab) Anti-TNF (infliximab)

Patients will be provided these medications as part of their standard of care, as decided by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ulcerative colitis who are beginning tofacitinib therapy.
2. Patients with ulcerative colitis who are initiating second line biologic therapy with ustekinumab
3. Patients with ulcerative colitis who are initiating second line biologic therapy with infliximab
4. Patients aged 18 years or older.
5. Patients with active disease defined as simple clinical colitis activity index (SCCAI) >2
6. Patients who have not been on antibiotics for 2 weeks or probiotics.

Exclusion Criteria:

1. Patients younger than 18 years.
2. Patients that do not meet the inclusion criteria specified above.
3. Patients with clinical signs of fulminant colitis, toxic megacolon, ischemic colitis or impending hospitalization for severe ulcerative colitis.
4. Patients with concomitant infectious colitis.
5. Patients allergic nuts/soy/sesame/oats.
6. Patients who do not like the food items that form part of the kits for the fasting mimicking diet (see below).
7. Patients that are diabetics on a glucose lowering drug.
8. Individuals with a history of syncope/presyncope with fasting or from medical conditions.
9. Women who are pregnant or nursing.
10. Individuals with very low BMI< or equal to 18.
11. Patients with the following comorbidities: chronic kidney disease, diabetes, active cancer.
12. Prohibited concomitant therapies will include TNF antagonists, azathioprine, methotrexate, and mercaptopurine.
13. Patients who routinely have fasting eating habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oriana Damas, MD, Principal Investigator — University of Miami
Locations (1):
- The University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data and code are available upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Advanced Therapy Plus FMD Group: Participants in this group with UC will start an advanced therapy with the addition of two, five-day cycles of Fast Mimicking Diet (FMD) daily meals on weeks 2 and 6.
  Fast Mimicking Diet: FMD is a five day meal plan that includes foods such as soups, snacks, bards, teas and supplements (omega-3 fatty acids) for a total of 66 items per box. The diet is plant-based, gluten free and dairy free without any artificial preservatives, chemicals or biologically active ingredients.
- Advanced Therapy Only Group (no Diet Intervention): Participants in this group with UC will initiate an advanced therapy and follow a diet based on dietary tolerances.
Period: Overall Study
Arm/Group | Advanced Therapy Plus FMD Group | Advanced Therapy Only Group (no Diet Intervention)
Started | 14 | 18
Completed | 9 | 12
Not Completed | 5 | 6
Not completed — Adverse Event | 2 | 0
Not completed — abdominal pain after starting tofacitinib | 1 | 1
Not completed — did not want to follow diet | 1 | 0
Not completed — flare up of ulcerative colitis | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — initiated another diet on their own | 0 | 2

BASELINE CHARACTERISTICS:
Population: This is the participant flow diagram of all patients inlcuded in the study and analyzed in the intention to treat arm.
Groups:
- Advanced Therapy Plus FMD Group: Participants in this group with UC will start an advanced therapy for eight consecutive weeks with the addition of two, five-day cycles of Fast Mimicking Diet (FMD) daily meals on weeks 2 and 7.
  Fast Mimicking Diet: FMD is a five day meal plan that includes foods such as soups, snacks, bards, teas and supplements (omega-3 fatty acids) for a total of 66 items per box. The diet is plant-based, gluten free and dairy free without any artificial preservatives, chemicals or biologically active ingredients.
- Advanced Therapy Only Group (no Diet Intervention): Participants in this group with UC will be begin an advanced therapy and consume a a diet based on dietary tolerance.
- Total: Total of all reporting groups
Arm/Group | Advanced Therapy Plus FMD Group | Advanced Therapy Only Group (no Diet Intervention) | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 29
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 25
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Simple clinical colitis activity index [Median (Inter-Quartile Range); unit: units on a scale] — SCCAI is a symptom-based questionnaire addressing five assessments, including bowel frequency day, bowel frequency night, urgency of defecation, blood in stool and general well-being. The SCCAI has a total range from 0-19 with a higher score indicating greater disease activity.
  units on a scale | 8.0 [6 to 12] | 7.0 [5 to 9] | 7.5 [5 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieved Clinical Response
Description: Clinical response will be evaluated using the Simple Clinical Colitis Activity Index (SCCAI). The SCCAI has a total range from 0-19 with a higher score indicating greater disease activity. A clinical response is defined as a SCCAI decrease of ≥3 points from baseline. Therefore, the study team will examine the percentage of patients who achieve 'clinical response', defined by an SCCAI decrease of ≥3 points.
Time Frame: 8 weeks
Measure: Number; unit: percentage of patients
Groups:
- Advanced Therapy Plus FMD Group: Participants in this group with UC will initiate an advanced therapy for UC for eight consecutive weeks with the addition of two, five-day cycles of Fast Mimicking Diet (FMD) daily meals on weeks 2 and 7.
  Type of advanced therapy is decided by the provider as part of the standard of care.
  Fast Mimicking Diet: FMD is a five day meal plan that includes foods such as soups, snacks, bards, teas and supplements (omega-3 fatty acids) for a total of 66 items per box. The diet is plant-based, gluten free and dairy free without any artificial preservatives, chemicals or biologically active ingredients.
- Advanced Therapy Without FMD (Medication Only Group): Participants in this group with UC will initiate an advanced therapy as their standard of care.
  Patients will be provided guidance on following a diet based on dietary tolerances.
Arm/Group | Advanced Therapy Plus FMD Group | Advanced Therapy Without FMD (Medication Only Group)
Number analyzed (Participants) | 14 | 18
percentage of patients | 57 | 35
Statistical Analysis 1: Comparison: Advanced Therapy Without FMD (Medication Only Group); Test type: Other; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Fecal Calprotectin Levels Measured in Micrograms/Gram
Description: Calprotectin levels were evaluated using fecal samples to compare the levels between the treatment and control arms before (baseline) and after the intervention (at 8 weeks). Fecal calprotectin was measured using a BUHLMANN fCAL ELISA Kit. Unit of measure was micrograms/gram.
Time Frame: baseline, 8 weeks
Measure: Mean (Full Range); unit: mcg/gram
Arm/Group | Advanced Therapy Plus FMD Group | Advanced Therapy Only Group (no Diet Intervention)
Number analyzed (Participants) | 3 | 5
mcg/gram
  Baseline | 3710 [456 to 30218] | 5138 [836 to 31594]
  Week 8 | 1375 [170 to 11197] | 5691 [926 to 34997]

3. Secondary Outcome: CRP Levels Measured in mg/dl
Description: Comparison of Median C-Reactive Protein (CRP) levels between the treatment and control arms before (baseline) and after the intervention (at 8 weeks) will be evaluated using blood samples, unit of measure was mg/dl
Time Frame: baseline, 8 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Advanced Therapy Plus FMD Group | Advanced Therapy Without FMD (Medication Only Group)
Number analyzed (Participants) | 6 | 6
mg/dl
  Baseline | 0.45 [0.33 to 0.73] | 2.10 [1.25 to 3.33]
  Week 8 | 0.09 [0.09 to 0.25] | 1.10 [0.53 to 2.73]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Any serious adverse event was reported to the sponsor of the study (Pfizer) and to the IRB. Pfizer funded this PI-initiated study.
  Non-serious events were recorded by our team and followed up on.
Groups:
- Advanced Therapy Plus FMD Group (Diet Intervention): Participants in this group with UC consuming a standard, regular low-fiber diet will start an advanced therapy for eight consecutive weeks with the addition of two, five-day cycles of Fast Mimicking Diet (FMD) daily meals on weeks 2 and 6.
  Medications started have been described previously.
  Fast Mimicking Diet: FMD is a five day meal plan that includes foods such as soups, snacks, bards, teas and supplements (omega-3 fatty acids) for a total of 66 items per box. The diet is plant-based, gluten free and dairy free without any artificial preservatives, chemicals or biologically active ingredients.
- Advanced Therapy Only Group (no Diet Intervention): Participants in this group with UC consuming a standard, regular low-fiber diet will be starting an advanced therapy (but not diet intervention).
  Medications started have been described previously.
Arm/Group | Advanced Therapy Plus FMD Group (Diet Intervention) | Advanced Therapy Only Group (no Diet Intervention)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/18
Other Adverse Events (participants affected / at risk) | 1/14 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Therapy Plus FMD Group (Diet Intervention) (N=14) | Advanced Therapy Only Group (no Diet Intervention) (N=18)
Hospitalization (Immune system disorders) | 2 (2) | 0 (0) — Both patients who had serious adverse events were admitted to the hospital for flares related to their disease condition (ulcerative colitis). Although both patients were in the intervention group, neither had initiated the dietary intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Therapy Plus FMD Group (Diet Intervention) (N=14) | Advanced Therapy Only Group (no Diet Intervention) (N=18)
abdominal pain (Immune system disorders) | 1 (1) | 2 (2) — 1. patient in the intervention arm had abdominal pain after initiating the advanced therapy (tofacitinib) and withdrew from the study. 2. patients in the control arm had abdominal pain after initiating the advanced therapy.

LIMITATIONS AND CAVEATS:
First, due to the COVID pandemic, we were unable to reach the recruitment numbers. Another limitation: initial protocol designed to only examine patients initiating tofacitinib but delays in recruitment due to COVID, together with the approval of upadacitinib, led to poor recruitment. Then expanded criteria to include: upadacitinib and to patients initiating their second- or third-line biologic (infliximab, ustekinumab, or risankizumab). Also sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT04505410/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04505410/ICF_001.pdf